CLINICAL TRIAL: NCT07241442
Title: Clinical Superiority of Cross-linked Hyaluronic Acid in Knee Osteoarthritis: Sustained Efficacy on Pain and Function
Brief Title: Cross-linked Hyaluronic Acid in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Seyda Ersahan, DDS, PhD, Assoc.Prof., Istanbul Medipol University Hospital
Other Study IDs: E-10840098-202.3.02-5817
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Knee Osteoarthritis, Cross-linked Hyaluronic Acid, Recreational Athletes, Intra-articular Injection, WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Straight-bonded hyaluronic acid — Straight-bonded HA injection was applied in 2 doses, 4 weeks apart.
Drug: cross-linked hyaluronic acid — Cross-linked HA was applied as a single dose to the knee via the anterolateral approach.

SUMMARY:
Knee Osteoarthritis (Knee OA) leads to pain and loss of function, especially in recreational athletes. While hyaluronic acid (HA) injections are a common part of conservative treatment, comparative data on the efficacy of straight-chain (ST-HA) versus cross-linked (CL-HA) formulations remain limited. Therefore, the aim of this study was to compare the 6-month efficacy of a single dose of CL-HA versus two doses of ST-HA regarding pain, stiffness, and joint function in recreational athletes aged 50-70 with Kellgren-Lawrence grade 2-3 Knee OA refractory to pharmacological treatment.

DETAILED DESCRIPTION:
This retrospective observational study included 88 recreational athletes (CL-HA: n=44, ST-HA: n=44). All participants received either a single dose of CL-HA or two doses of ST-HA administered 4 weeks apart. Patients were comparatively evaluated pre-treatment and at 1, 3, and 6 months post-treatment using the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) and VAS scores.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria: Recreational athletes aged 50-70 years; participants must not have received any injections or undergone physical therapy or rehabilitation in the last 3 months; and symptomatic cases of Kellgren-Lawrence stage 2-3 knee osteoarthritis and failure of pharmacological treatment.

Exclusion Criteria: Inflammatory disease, active rheumatic disease, malignancy, bleeding diathesis, peripheral neuropathy, BMI >30, grade 4 gonarthrosis, regular NSAID use, previous knee surgery, local infection at the procedure site, corticosteroid injection at the procedure site within the last 3 months, systemic corticosteroid use within the last 2 weeks, immunosuppressant use or immunodeficiency within the last 6 weeks, and any local or systemic osteoarthritis-related treatments (therapeutic exercises, physical therapy, other injections, NSAIDs, etc.) within the last 6 months.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective observational study was conducted in a multicenter manner and included recreational athletes aged between 50 and 70 years who applied to Medipol Esenler Hospital and Republic of Turkey Ministry of Health Erenköy Physical Therapy and Rehabilitation Hospital due to knee pain and were diagnosed with gonarthrosis between January 2021 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Patients were comparatively evaluated pre-treatment and at 1, 3, and 6 months post-treatment using the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score. | Patients were comparatively evaluated pre-treatment and at 1, 3, and 6 months post-treatment

SECONDARY OUTCOMES:
Patients were comparatively evaluated pre-treatment and at 1, 3, and 6 months post-treatment using the VAS score. | Patients were comparatively evaluated pre-treatment and at 1, 3, and 6 months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After publication in a journal, I will share all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning immediately after publicaiton
Access Criteria: I will consider review requests for IPD sharing and how they will be reviewed.